CLINICAL TRIAL: NCT02247778
Title: Outcome of Mini-incision-technique for Treatment of Midshaft Fractures of the Clavicle
Brief Title: Surgical Innovations in Treatment of Clavicle Fractures
Acronym: ClavFrac
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Chlodwig Kirchhoff, PD DR. med. Chlodwig Kirchhoff, Technical University of Munich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beiromat_02
Record Dates: First submitted 2014-09-21; First posted 2014-09-25 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Complication
Keywords: clavicle; surgical intervention; mini-incision; plate osteosynthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional plate osteosynthesis (Active Comparator): Standard procedure
  Interventions: Procedure: conventional plate osteosynthesis
- mini-incision-type osteosynthesis (Active Comparator): mini-incision
  Interventions: Procedure: mini-incision-type osteosynthesis

INTERVENTIONS:
Procedure: conventional plate osteosynthesis — Standard incision
  Arms: conventional plate osteosynthesis
Procedure: mini-incision-type osteosynthesis — Mini-incision
  Arms: mini-incision-type osteosynthesis

SUMMARY:
Surgical incision for plate osteosynthesis of midshaft fractures of the clavicle averages 7 to 8 centimeters in the literature. It is hypothesized, that depending on the invasiveness of this incision secondary problems like prolonged fracture healing, paresthesia of supraclavicular nerves and pain due to scar tissue increase. Therefore we developed a mini-incision technique using an average incision length of 4cm.

The aim of this study is to analyzed whether secondary problems following plate osteosynthesis of the clavicle correlate mit the length of the surgical access.

DETAILED DESCRIPTION:
Surgical incision for plate osteosynthesis of midshaft fractures of the clavicle averages 7 to 8 centimeters in the literature. It is hypothesized, that depending on the invasiveness of this incision secondary problems like prolonged fracture healing, paresthesia of supraclavicular nerves and pain due to scar tissue increase. Therefore we developed a mini-incision technique using an average incision length of 4cm.

The aim of this study is to analyzed whether secondary problems following plate osteosynthesis of the clavicle correlate mit the length of the surgical access. Therefore a prospective observational protocol was chosen.

ELIGIBILITY:
Inclusion Criteria:

all patients with fractures of the clavicle and indication for operative intervention using plate osteosynthesis ability to sign informed consent

Exclusion Criteria:

all other patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
area of paresthetic skin | 12 month

SECONDARY OUTCOMES:
Time to fracture healing | 12 month
Postoperative shoulder function | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Chlodwig Kirchhoff, MD, Principal Investigator — Klinik und Poliklinik für Unfallchirurgie, Klinikum rechts der Isar, Technische Universität München
Locations (1):
- Klinik und Poliklinik für Unfallchirurgie, Klinikum rechts der Isar, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Beirer M, Postl L, Cronlein M, Siebenlist S, Huber-Wagner S, Braun KF, Biberthaler P, Kirchhoff C. Does a minimal invasive approach reduce anterior chest wall numbness and postoperative pain in plate fixation of clavicle fractures? BMC Musculoskelet Disord. 2015 May 28;16:128. doi: 10.1186/s12891-015-0592-4. PMID 26018526